CLINICAL TRIAL: NCT04453293
Title: A Proof-of Concept, Randomized, Controlled Study of Tuberculosis Immunization With BCG to Prevent Infection in Healthy Adults (TIPI Trial)
Brief Title: Immunization With BCG Vaccine to Prevent Tuberculosis Infection
Acronym: TIPI
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The sponsor has elected to discontinue/terminate the study prematurely due to slower-than-anticipated recruitment and limited remaining research funding.
Sponsor: Henry M. Jackson Foundation for the Advancement of Military Medicine (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2019-01; BAA 170090 (Other Grant/Funding Number: Defense Health Program (admin by MIDRP))
Record Dates: First submitted 2020-06-17; First posted 2020-07-01 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Tuberculosis Infection
Keywords: BCG Vaccine; Tuberculosis vaccine
MeSH Terms: conditions — Latent Tuberculosis | interventions — Vaccines; Sodium Glutamate

STUDY DESIGN:
Intervention Model Description: Randomized, controlled trial of BCG (Tokyo 172) vaccine single dose given intradermally compared to placebo vaccine (diluent) given intradermally single dose
Who Masked: Participant
Masking Description: The participant and the laboratory (endpoint measurement) will be masked
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BCG vaccine (Experimental): Freeze-dried Glutamate Bacillus Calmette-Guérin (BCG) (Tokyo 172) vaccine
  Interventions: Biological: BCG (Tokyo 172) vaccine
- Placebo (Placebo Comparator): Vaccine diluent [sodium glutamate]
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: BCG (Tokyo 172) vaccine — Freeze-Dried Glutamate Bacillus Calmette-Guérin BCG Vaccine (Japan BCG Laboratory), 0.1 mL given as single dose by intradermal injection over the outer lower aspect of the deltoid region
  Arms: BCG vaccine
Drug: Placebo — Placebo vaccine diluent, 0.1 mL given as single dose by intradermal injection over the outer lower aspect of the deltoid region
  Other Names: sodium glutamate
  Arms: Placebo

SUMMARY:
The purpose of this research is to find out if a single dose of pre-travel vaccination with BCG can lessen tuberculosis (TB) infection by producing an immune response when given to adults traveling to countries with a high or moderate burden of TB. BCG will be compared with a placebo (an inactive vaccine). BCG (Japan) is used globally but is not approved for use in the United States, therefore it is considered experimental. Participants choosing to take part in this research study, will be randomly assigned (this is like a coin flip) to BCG or placebo. 2000 eligible volunteers will be enrolled.

DETAILED DESCRIPTION:
This study is a multi-center, prospective, randomized, placebo-controlled, participant and laboratory-blinded clinical trial to evaluate a single pre-travel vaccination with investigational freeze-dried glutamate BCG (Japan) to prevent Mycobacterium tuberculosis complex (Mtb) infection in healthy adult travelers, 18-65 years of age, exposed to persons with TB in high or moderate burden countries.

The goals of this study are both public health and scientific. The public health goal of this study is to offer possible protection against TB to US workers traveling abroad to work in countries with a high burden of TB where there is a risk for multidrug resistant/extensively drug resistant TB exposure and where effective TB infection control interventions are infrequently fully implemented. A long-term scientific goal is to test the hypothesis that TB vaccination prevents primary TB infection as measured by peripheral blood TB interferon gamma release assay (IGRA) conversion at return from travel visit, as well as sustained conversion at approximately 4-6 months post-return from travel. Rates of IGRA conversion in BCG-vaccinated recipients as compared to placebo recipients will be evaluated. Additionally, this study will collect information regarding exposure to and infection with TB, assessing risk factors for TB infection during the participant's travel.

This study will recruit health care workers (public health workers or students in training status) traveling to countries with a high or moderate burden of TB where there is a risk for multidrug resistant/extensively drug resistant (MDR/XDR) for a minimum of 10 days up through 6 months, with planned exposure to the local population such as patient care activities. Performance sites will not enroll anyone traveling for greater than 6 months or longer.

High or moderate TB burden countries for this study are defined as countries identified in the World Health Organization (WHO) Global Tuberculosis Report 2020 to have a TB incidence of ≥20/100,000. Targeted participant population of travelers at-risk for high TB exposure will work specifically in one or more of the 131 highest ranked TB burden countries as recognized by the WHO 2020 report.

Participants enrolled will be required to complete typically 4, but up to 6 study visits composed of: screening and eligibility assessments, vaccination with study vaccine (BCG or placebo), a subsequent post-vaccination follow-up assessment visit to identify potential adverse event occurrences, a post-travel follow-up visit to assess the risk factors for Mtb infection and assess the primary endpoint (IGRA conversion from negative to positive), and if applicable, an additional visit for those participants who are found to have a borderline IGRA result. For participants found to have post-travel IGRA conversion results, an additional visit will be requested for assessment of sustained TB IGRA conversion and reversion.

Different evaluations, tests and/or procedures to be performed during study visits include: interviews relevant to their medical history and general well-being between study visits; physical examinations and vital signs; completion of a pre-travel questionnaire and post-travel questionnaires to collect information regarding exposure to TB and risk factors for infection, as well as any information regarding development of active TB disease, both pulmonary and/or extrapulmonary and evaluation for the presence and severity of self-reported symptomatic all-cause respiratory infection occurrences while traveling abroad; keeping a record to assess for occurrence of local reactions at the injection site and incidence of selected symptoms for the first 14 days post-vaccination; and blood draws (2 up to 4 depending on what previous blood test results reveal).

The study design is endpoint driven; designed to observe 56 total IGRA conversions. Therefore, enrollment into this study will be stopped if the target endpoint (56 IGRA conversions) are met earlier than expected.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be eligible for study participation if they meet all of the following criteria:

  1. Participant is willing to participate in the study as evidenced by providing voluntary written informed consent and Health Insurance Portability and Accountability Act (HIPAA) authorization prior to conducting any trial related procedures
  2. Participant is male or female, age ≥ 18 years and ≤ 65 years at time of consent
  3. Participant is in good general health, confirmed by medical history, laboratory screening, and physical examination
  4. Participant has no known history of Mtb infection
  5. Participant has no prior history of BCG vaccination, or previous receipt of an investigational Mtb vaccine
  6. Participant is assessed to be at risk for TB exposure (particularly drug resistant TB) during planned travel and has planned to work in high or moderate TB burden countries for a duration of a minimum of 10 days and not greater than 6 months for HCW
  7. Participant presents at least 4 weeks prior to travel departure
  8. Participant is willing to forego any periodic tuberculin skin test screening procedures for 6 months after receiving BCG/placebo vaccine
  9. Participant is willing to wait after receiving a COVID-19 vaccine for 7 days before receiving BCG/placebo vaccine
  10. Participant is willing to complete all study visits as required by the protocol and is reachable by telephone or email during the study
  11. Participant agrees to medical record access for purposes of relevant medical history collection

      For Females of Childbearing Potential Only:
  12. Participant has a negative urine pregnancy test prior to starting study treatment
  13. Participant is willing to use effective contraception for at least 30 days before and 6 weeks after BCG/placebo vaccination
  14. Lactating female that is willing to refrain from breast-feeding for 6 weeks post-vaccination

Exclusion Criteria:

* Participants will be ineligible for study participation if they meet any of the following criteria:

  1. Participant has known positive tuberculin skin test (>10 mm) or positive IGRA
  2. Participant has medical condition for which BCG vaccination is contraindicated (e.g., HIV or other immunocompromised conditions)
  3. Participant is currently receiving (within last 30 days) immune-compromising treatments, such as TNF-α blockade
  4. Participant has history of chronic (≥ 30 days) oral steroid use or intravenous (IV) steroids within the last 90 days
  5. Participant has received radiation therapy or chemotherapy within the last 180 days
  6. Participant has received BCG treatment for bladder cancer
  7. Participant is female and is pregnant (as defined by positive urine βHCG test) or intends to become pregnant in next 3 months, or is breast-feeding at screening or vaccination visit
  8. Participant is unwilling to complete all required study elements (e.g., HIV testing)
  9. Participant has received 2 or more live vaccinations (e.g., measles and yellow fever) within 30 days prior to receipt of BCG/placebo vaccine (Visit 2)
  10. Participant has known or suspected hypersensitivity to BCG vaccine or related products
  11. Participant has positive/borderline IGRA test at screening
  12. Participant has positive/indeterminate HIV test at screening unless has received prior HIV vaccine
  13. Participant has a history of life-threatening adverse event following receipt of any immunization
  14. Participant is known to have a behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the participant to understand or cooperate with the requirements of the study protocol
  15. Participant has other concurrent condition(s) that in the opinion of the investigator would jeopardize the safety or rights of a participant participating in the trial or would render the participant unable to comply with the protocol and/or compromise study objectives
  16. Participant has had tuberculin skin testing performed within 1 month prior to Visit 1
  17. Participant has received a COVID-19 vaccine within 7 days prior to BCG/placebo vaccine
  18. Participant has had a probable exposure to TB (defined as to someone with suspected or confirmed pulmonary TB who is likely infectious) within 8-10 weeks of Visit 1
  19. Participant has prior history of nontuberculous mycobacterial disease, not colonization only

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2026-01-16 (Actual); Study Completion 2026-01-16 (Actual)

PRIMARY OUTCOMES:
Change in TB IGRA blood test results from baseline pre-travel and post-travel return | At baseline, and 8-10 weeks post-travel return
  Conversion change of TB IGRA from pre-travel baseline value of negative to positive post-travel, using FDA-approved breakpoints as a measure of Mycobacterium tuberculosis infection. Response will be assessed using technology of the T-SPOT.TB test method. Specifically, the test measures the number of spots from T cells sensitized to TB infection on a plate containing 4 different antigens: nil (negative control), 2 TB antigens (ESAT-6 and CFP-10, also called Panel A and Panel B), and phytohemagglutinin (positive control). Results are interpreted by subtracting the spot count in the negative (NIL) control from the spot count in Panels A and B:
  * Positive ≥ 8 spots
  * Negative ≤ 4 spots (this includes values less than zero)
  * Borderline 5, 6, or 7 spots
  * Invalid

SECONDARY OUTCOMES:
Number of Participants with sustained conversion and reversion in the TB IGRA converters | 4-6 months from return post-travel
  Participants identified as having positive TB IGRA blood test results will undergo a TB IGRA re-test to determine sustained (positive result) conversion and reversion (defined as negative/borderline) using the T-SPOT.TB test method. The rate of conversion for each study group will be calculated as the number of conversions divided by person-months of travel
Number of Participants with history of TB disease/symptoms while deployed | Through final IGRA testing, expected average time 8-10 weeks post-travel return
  Participants with response of symptoms suggestive of TB disease (i.e., bloody cough, cough ≥ 2 weeks, chest pain, fever ≥ 2 weeks, night sweats, and unintentional weight loss), development of active TB disease (possible, probable, or definite) and TB treatment that may have occurred during travel to high or moderate burden TB country or up to the time of IGRA testing.
Identify potential risk factors for Mtb infection in the targeted study population collected on Post-Travel Questionnaire | Through final IGRA testing, expected average time 8-10 weeks post-travel return
  Questionnaire responses from participants after travel will collect information regarding exposure to TB and risk factors for infection, as well as any information regarding risk reduction activities taken (i.e. personal protective measures) that may have occurred during travel to countries with high burden TB identified in the 2020 World Health Organization (WHO) TB report. Travelers will be asked if they had contact with anyone known to have TB disease or if they worked with populations at risk for HIV while abroad. They will also be asked about accommodations, daily routine, and if they used public transportation such as mini-buses and if so, how frequently. A final open-ended question e.g., "Do you have reason to believe you were exposed?" will be asked of all travelers
Number of Participants with treatment-related adverse effects following intradermal administration of BCG vaccine | Baseline (pre-administration of vaccine), within 30 minutes of vaccination, 14-days post-vaccination, and 2 to 6 weeks post-vaccination (Visit 3)
  Post-vaccination response to assess for occurrence of selected local injection site reactions (pain/tenderness, redness, ulceration, drainage, vesicle [blister], induration [swelling] and scarring), axillary/ cervical lymphadenopathy, and selected systemic symptoms (fever, headache, chills, dizziness, tiredness, nausea, gastrointestinal problems, rash, muscle and joint pain and general well-being) using the 2007 U.S. FDA guidance Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials. For each reaction, the highest grade will be determined for each traveler. Participants will be provided with a memory aid card to record any occurrences of selected local reactions and systemic symptoms that may occur during the first 14-days post-vaccination
Number of Participants with self-reported symptoms of all-cause respiratory infections acquired while traveling abroad | Through final IGRA testing, expected average time 8-10 weeks post-travel return
  Questionnaire responses obtained from participants will assess self-reported symptomatic all-cause respiratory infection symptoms in five domains (nose, throat, chest, systemic, neurological) for presence, frequency of occurrence and severity, impact of acute symptoms on functional activities or productivity, and medical care encounters and treatment as a result of respiratory illness while traveling abroad.

CONTACTS AND LOCATIONS:
Overall Officials: Naomi E. Aronson, MD, Study Chair — Uniformed Services University of the Health Sciences; Merlin L. Robb, MD, Study Director — Henry M. Jackson Foundation for the Advancement of Military Medicine
Locations (7):
- United States (7):
  - Yale University School of Medicine, New Haven, Connecticut
  - MedStar Washington Hospital Center/MedStar Health Research Institute, Washington D.C., District of Columbia
  - Hope Clinic of the Emory University Vaccine Center, Emory University, Decatur, Georgia
  - Johns Hopkins Bloomberg School of Public Health, Department of International Health, Center for Immunization Research, Baltimore, Maryland
  - The Brigham and Women's Hospital Center for Clinical Investigation, Boston, Massachusetts
  - Baylor College of Medicine, Houston, Texas
  - University of Utah School of Medicine, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2021-09-22): https://cdn.clinicaltrials.gov/large-docs/93/NCT04453293/ICF_001.pdf